CLINICAL TRIAL: NCT01550640
Title: Pharmacogenetics of Remifentanil in Patients With Hypertension Undergoing Cesarean Delivery Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: General Teaching Hospital, Prague (Other)
Responsible Party: Principal Investigator, Jan Blaha, MD, PhD., Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: remifentanil
Record Dates: First submitted 2012-03-06; First posted 2012-03-12 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy; Cesarean Delivery; General Anesthesia
Keywords: remifentanil; Caesarean operation; general anaesthesia; hypertension; newborn's adaptation; pharmacogenetics
MeSH Terms: conditions — Hypertension | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- remifentanil (Experimental): bolus of remifentanil 1 µg/kg will be given 30 sec before induction to general anesthesia
  Interventions: Drug: Remifentanil
- standard (No Intervention): control standard group

INTERVENTIONS:
Drug: Remifentanil — bolus of remifentanil 1 µg/kg will be given 30 sec before induction to general anesthesia
  Other Names: Ultiva
  Arms: remifentanil

SUMMARY:
Caesarean delivery under general anaesthesia (GA) carries nowadays still 25% risk of insufficient depth of anaesthesia in a time before the fetus delivery. The reason is the lack of opioid administration. Opioids easily cross placental barrier and negatively influence newborn postpartum adaptation by respiratory depression. Introduction to GA is thus accompanied by exaggerated autonomic stress reaction with hypertension and tachycardia. The use of ultra-short acting opioid remifentanil should suppress stress response in mother without increasing the risk for newborn. There are only a few clinical data available. This study will be the first one systematically studying the influence of remifentanil in pregnant women with hypertension on hemodynamic stability and newborns safety. This study will also identify potential pharmacogenetic factors of individual variability in remifentanil response with respect of drug efficacy and safety in mother and newborn.

DETAILED DESCRIPTION:
INTRODUCTION Even nowadays there is still a significant risk of insufficient depth of anesthesia during Cesarean delivery (CD) under general anesthesia (GA). The main reason in comparison to other surgeries is the lack of opioid administration due to risk of newborn respiratory depression.

Opioids easily cross the placental barrier to the fetus circulation and may cause depression of respiration and deteriorate the overall newborns postpartum adaptation. This presents the main reason why according to contemporary recommendation is the use of opioids in CD restricted until the time of fetus delivery, and are given as far as after the navel wort ligation. Not to cause any depression of the newborn the premedication to GA is usually also omitted. The beginning of GA in common surgical operation is usually accompanied by the decrease in systemic blood pressure (BP) and heart rate (HR). However, in CD the investigators face the increase of BP and HR due to stress reaction of mother during the period before the fetus delivery and before full anesthesia application, including opioids.

Generally, insufficient depth of anesthesia (assessed by patient's recollection) is reported in less than 1% of cases, but increases for up to 50% in GA during CD. However, this appraisal marginalized much more frequent cases when an insufficient depth of GA is accompanied by exaggerated autonomic reaction to the pain, especially the increase in systemic BP and heart rate as a reaction to the egestion of catecholamines, while total amnesia of the surgery is retained. In CD such type of anesthesia insufficiency was reported in 12-26% of patients! Current trend in CD anesthesia unequivocally prefers the use of regional techniques; GA remains indicated for emergency situations mainly and in those cases the stress reaction of mother tends to be much higher than in elective procedures.

An independent remarkable risk factor to the pregnant women is the hypertension, both chronic and gestational including preeclampsia. This condition of preoperatively mostly hardly and insufficiently controlled hypertension may get dramatically worse during the first phase of CD, when blood pressure due to uncontrolled stress reaction enormously rises and elevates intracranial pressure with high risk of hemorrhagic stroke - a life threatening complication.

Unfortunately there are only a few possibilities how to influence mother's stress response to intubation and laparotomy without increasing the risk of newborn depression. In absence of anesthetics not crossing placental barrier, the only possibility is the use of ultra-short acting anesthetics which should be eliminated from fetus circulation before his delivery. An important role might play remifentanil - µ-receptor agonist with rapid onset and ultra-short activity (biological half-life 3-10 min.). It's major advantage, beside fast onset, is also prompt and organs independent elimination.

HYPOTHESIS Bolus administration of an ultra-short acting synthetic µ-opioid receptor agonist, remifentanil, in mothers with hypertension/preeclampsia before induction of general anesthesia attenuates egestion of stress catecholamines and development of stress autonomic reaction in response to laryngoscopy, intubation and subsequent laparotomy during CD. The remifentanil administration thus suppress the hypertensive and tachycardiac increase during the initial period of CD , but without negative influence on newborns postpartum adaptation, mainly breathing. On the contrary the prevention of uteroplacental blood flow reduction should improve the postpartum adaptation of the newborn. The project should also give pilot data, if genetic polymorphisms of target genes, important for remifentanil pharmacokinetic and pharmacodynamic, influence in Czech population drug efficacy and safety.

As extrapolated result the investigators expect the reduction of complications attributed to severe BP increase, especially hemorrhagic stroke. The remifentanil administration should not have any negative influence on newborn, especially on postnatal adaptation and breathing activity. Prevention of uteroplacental insufficiency in response to hypertension and tachycardia may even lead to better newborn status.

AIMS

The aims of the project are:

1. To assess newborn postnatal adaptation after cesarean delivery under general anesthesia with a remifentanil bolus 1 µg/kg prior to the induction of general anesthesia
2. To demonstrate a stabilizing influence of remifentanil on circulation and depth of anesthesia in patients with hypertension/preeclampsia in the time of fetus delivery during CD
3. To assess the influence of individual hereditary variability in MDR1 (multidrug resistance gene 1) and PXR (pregnane X receptor) on RMF pharmacodynamics.
4. To assess the influence of individual genetic variability in µ-opioid receptor gene on drug effects in newborn.

Extrapolated result should be both the reduction of complications in mother associated with serious increase in systemic blood pressure and improved postpartum newborn adaptation. Patients with hypertension/preeclampsia are at high risk of insufficient depth of anesthesia during CD and this may lead to uncontrolled hypertension with the risk of intracranial bleeding. To avoid this complication represents one of current obstetrician anesthesia priorities. Optimal introduction to GA in this clinical situation has not been yet identified.

METHODS AND RESEARCH SAMPLE Type of study: prospective, randomized, double-blinded for the assessment of neonatal adaptation and single-blinded for the evaluation of haemodynamic changes.

Patient file: 160 pregnant women undergoing CD under GA; 80 patients with hypertension/preeclampsia - 40 in the REMIFENTANIL group and 40 in the STANDARD (placebo) group; 80 patients without hypertension/preeclampsia - 40 in the REMIFENTANIL group and 40 in the STANDARD (placebo) group.

Randomization: Will be performed before CD using the envelope method. Randomization and preparation the appropriate study bolus (remifentanil 1 µg/kg) will be performed by supervising anesthesiologist. The randomization for the neonatologist will be broken in the case of medical complication, e.g. when respiratory depression in infant occurs and opioid antagonist may be administered. Supervising anesthesiologist will not otherwise interfere with the course of CD or evaluation of the data.

Conduct of anesthesia: Thirty seconds prior to GA induction bolus of study drug solution is given intravenously. Afterwards anesthesia will be conducted in a standard way: induction to GA with combination of thiopentone 5 mg/kg and suxamethonium 1.25 mg/kg; subsequent intubation and inhalation of oxygen/nitrous oxide (1:1) and sevoflurane 0.7%. Following the intubation neuromuscular relaxant Atracurium is administered 0.35 mg/kg. After delivery of the newborn and umbilical cord clamping opioid analgesia with sufentanil 0.3-0.5 µg/kg and inhalation of oxygen/nitrous oxide (2:3) + sevoflurane 0.7-1.0% will be administered. If required, additional bolus of sufentanil 10 µg intravenously will be given.

Intraoperative monitoring: All the patients will be monitored according to guidelines with respect to risk associated with hypertension/preeclampsia and GA for CD - ECG (including V4-5 thoracic lead, ST analysis), SatO2, ETCO2, % of oxygen, % of volatile anesthetics, ventilation parameters (PIP, MV, TV, F).

For evaluation of anesthesia depth continuous bispectral EEG analysis (BIS) and sympathetic skin reflex response (SSRR) will be used. BIS is electrophysiological method reflecting the inability to perceive stimuli from environment using mathematical analysis of EEG curve; SSRR is unique method measures changes of skin conductivity that with high sensitivity and delay of only 1-2 sec. reflects immediate changes in sympathetic system to nociceptive stimuli (Stress Detector; Med-Storm, Norway).

DATA COLLECTION Demographics: age, height, weight, BMI, gestational age, previous pregnancy, associated medical conditions.

Preoperative laboratory values (haematology, liver and kidney function, total protein). Hemodynamics (BP, MAP, HR, ST analysis), ventilation (MV, SatO2, ETCO2), depth of anaesthesia (BIS, SSRR). Time course of CD (study drug administration, induction to GA, intubation, beginning of surgery, hysterotomy, delivery). Measurement of blood loss, complications.

Clinical examination and assessment of newborn status (Apgar score + acid-base measurement from umbilical cord, clinical evaluation and scoring).

Biological material sampling To assess genotype of MDR1 gene and PXR (Pregnane X Receptor) 8 ml of umbilical blood and 8 ml of venous blood from mother will be collected.

Pharmacogenomic analysis: Validated methods for PXR and MDR1 polymorphism analysis are available at our workplace. In both genes five polymorphisms with possible functional impact will be analyzed in every sample. Method for assessment of opioid receptor polymorphism (A118G) will be implemented during the first year of the study.

EVALUATION Level of anesthesia depth will be evaluated by BIS and SSRR values and by hemodynamic response to intubation and incision, especially by changes of BP (systolic, diastolic, mean) and heart rate.

Evaluation of newborn status will be assessed by Apgar score and acid-basis measurement of umbilical cord blood and by clinical assessment and scoring performed by experienced neonatologist.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women,
* age 18-45
* Cesarean delivery under general anesthesia
* informed consent

Exclusion Criteria:

* non-cooperative patient
* previous allergy to remifentanil or additional substance
* multiparity
* age of foetus <35th week
* estimated foetus weight <2500 g
* hypoxia or other signs of foetus distress
* mother's hypotension

Discontinuation Criteria:

- difficult foetus delivery (uterine incision-to-delivery interval >3 min)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Newborn adaptation after delivery | 10 min after delivery
  newborn status (Apgar score + acid-base measurement from umbilical cord, clinical evaluation and scoring)
Influence of individual hereditary variability in MDR1 (multidrug resistance gene 1) and PXR (pregnane X receptor) on remifentanil pharmacodynamics. | at time of delivery

SECONDARY OUTCOMES:
Depth of anesthesia | 30 min from induction to general anesthesia
  BIS (continuous bispectral EEG analysis)
Hemodynamic response to intubation and beginning of Cesarean operation | 30 min from induction to general anesthesia
  Changes in major hemodynamic parameters (Systolic Blood Pressure, Heart Rate, ST analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Blaha, MD, PhD., Principal Investigator — General University Hospital, Prague
Locations (1):
- General University Hospital in Prague, Prague, Czechia

REFERENCES:
- [Derived] Noskova P, Blaha J, Bakhouche H, Kubatova J, Ulrichova J, Marusicova P, Smisek J, Parizek A, Slanar O, Michalek P. Neonatal effect of remifentanil in general anaesthesia for caesarean section: a randomized trial. BMC Anesthesiol. 2015 Mar 26;15:38. doi: 10.1186/s12871-015-0020-1. eCollection 2015. PMID 25821405